CLINICAL TRIAL: NCT03261076
Title: Severe LD in Juvenile Delinquents: Presentation, Course, and Remediation
Brief Title: Reading Remediation and Outcomes in Detention
Acronym: SERIOUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Houston (Other); Harris County Juvenile Probation Department (Unknown); Connecticut Court Support Services Division (Unknown); MindTrust Labs (Unknown)
Responsible Party: Principal Investigator, Elena, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-40232
Record Dates: First submitted 2017-07-21; First posted 2017-08-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Specific Learning Disorder (MeSH Unique ID: D000067559); Dyslexia (MeSH Unique ID: D004410); Conduct Disorder (MeSH Unique ID: D019955)
Keywords: Specific Learning Disorder; Learning Disorders; Neurodevelopmental Disorders; Mental Disorders; Developmental Reading Disability; Reading Disorder; Conduct Disorder
MeSH Terms: conditions — Specific Learning Disorder; Dyslexia; Conduct Disorder; Learning Disabilities; Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a multiple baseline design, in which participants enter into the single-arm intervention at different times, yet have data collected at all time points. Approximately one third of participants will have their entry into the intervention shifted later by one week, and approximately another third will have their entry shifted by two weeks. This will happen on a rotating basis. All individuals will receive progress monitoring during the weeks that the other individuals are receiving intervention and/or assessments. The multiple baseline design allows for all individuals to receive the study intervention, and still provides a mechanism for monitoring change (or lack thereof) during non-intervention periods before and after intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SERIOUS Intervention (Experimental): All youth will be juveniles in a residential facility for post-adjudicated youth. They will be recruited into the study as they are being placed in the facility post-adjudication, to ensure that they meet criteria and will be in the facility long enough to complete the program. All qualified youth will be invited to participate in the SERIOUS intervention; once a group of youth are recruited to complete the multiple baseline design and interventionists are free (from running interventions with other participants) to work with the youth, an intervention cycle will begin.
  Interventions: Behavioral: Strategies Enhancing Reading in Older Underperf. Students

INTERVENTIONS:
Behavioral: Strategies Enhancing Reading in Older Underperf. Students — Strategies for Enhancing Reading in Older Underperf. Students (SERIOUS) combines two scientific, research based intervention programs, each meeting specific need of youth in detention: (1) Stevenson Reading Program, manualized and uniquely suited to students with phonological awareness, attention, and memory difficulties that may impact reading; and (2) Dr. Sharon Vaughn's well-documented, validated program, explicitly designed for older, severely reading-impaired students. SERIOUS also includes: (3) metacognitive strategies for self-regulated learning, and (4) A gamified extension of the intervention on a SmartPhone, designed to reinforce word-level skills (e.g., decoding, automaticity, and vocabulary), and including features efficacious for learning.

SUMMARY:
The current literature on academic skill difficulties, whether considered as part of the continuum of ability or as a specific learning disability (LD), indicates that these problems often coexist with conduct problems and juvenile delinquency, and are risk factors for initial law-breaking behavior and for its persistence. However, less is understood about how this relationship develops. It is these broad questions that this project seeks to address. First, what is the causal pathway? Does LD cause delinquency, delinquency cause LD, or are both caused by something else? And can big data analytics applied to statewide datasets of information about juvenile justice (JJ) involvement help to answer this question? Second, as it is known that learning to read and do math (and thus becoming more employable) increases the likelihood of desistance (i.e., not committing any more illegal acts), what are the necessary parts of an intervention designed to teach these skills? And what role might technology play in such an intervention? To answer these questions, we will implement a study that includes two components, (a) a big data component and (b) an intervention component. For (a), we will work with a large historical dataset from the Harris County Juvenile Probation Department. For (b), we will work, in total, with 192 (48 per year) delinquent youth with severe LD in residential placement. These individuals, in a nonconcurrent multiple baseline design, will be offered an educational therapy designed to address severe reading problems in juvenile detainees using a novel mixed media intervention in which the person-to-person intensive 1:1 component is completed while youth are in residential settings (24 sessions, delivered in 90 minute settings 3 times a week) and a "gamified" educational smartphone learning tool follow-up completed upon release (with appropriate network fidelity monitoring and participant reinforcement). The person-to-person component is developed specifically for juvenile offenders with severe LD, combining two well-established and highly-regarded intervention programs designed to systematically build students' repertoire of grapheme-phoneme correspondence rules as well as develop comprehensive reading skills, from beginning reading to proficiency.

DETAILED DESCRIPTION:
Learning disabilities (LD) are among the most common types of disabilities in juvenile offenders that have been linked to delinquency. Nationwide, children and youth with special education needs are overrepresented in the US justice systems. Reports estimate delinquent juveniles with a disability to comprise about 30% to 60% of the entire delinquent population. A national survey in the US states an average prevalence rate of 33.4% of incarcerated juveniles with disabilities in correctional facilities. Moreover, concerns have long been raised on the recidivism rates of youth with disabilities and special education backgrounds. In general, regarding educational performance, academic deficits such as a lack of basic skills in reading, writing, and mathematics have been associated with recidivism. However, these studies largely neglect the dynamic nature of delinquent and criminal behavior that has been documented within the field of developmental criminology with a focus on the onset, continuity, and extinction of deviant behavior. In light of this research, the identification and remediation of LD as a risk factor for repeat offending has been a persistent challenge given the accumulation of and overlap with other risk factors such as poverty, familial patterns of criminality, influence of delinquent peers, and the differential impact of risk factors across an individual's developmental trajectory. Altogether, there is a challenge around the implementation of sophisticated methodology to model the complex longitudinal and reciprocal links between juvenile delinquency and educational problems such as LD, and how they relate to other risk factors over time. This challenge is intensified by the required large samples to detect robust and interpretable patterns and predictive relationships for groups of youth with severe LDs that, by definition, are small in size and censored with regard to various educational outcomes (e.g., academic performance). This research is conceived to contribute to the field's understanding of the connection between LD and delinquent behavior. We hope to generate unique findings capitalizing on the availability of the relevant big data, the clinical strengths of its members and their capacity to develop and administer educational therapy to juvenile offenders, and its embedment within communities empowering the creation and processing of multi-level longitudinal datasets, merging sociological (i.e., criminological), behavioral, neurophysiological, and genetic/genomic data.

Big Data:

The Big Data component seeks to address three objectives: (1) to conduct big data analytics and data mining to quantify/qualify the complexities of severe LD among juvenile justice (JJ)-involved youth using statistical methods applied to big datasets that capture multiple indicators (i.e., offending and educational outcomes) cross-sectionally (for one-time offenders) and longitudinally (for repeat offenders); (2) to utilize big data analytics to identify a group of youth with severe LD who will serve as a comparison group for individuals participating in a reading intervention; and (3) to evaluate the findings from the first two objectives based on the statistical assumptions underlying the models applicable to the big data at hand.

Hypotheses. Extending previous research, Big Data seeks to identify factors that relate LD to recidivism, frequency of re-offending and re-arrest, and the time to post-involvement recidivism. We hypothesize that (a) overall recidivism rates (i.e., regardless of the specific type of offense) will be higher among JJ-involved youth with severe LD (operationalization based on standardized achievement tests and special education status) than in youth without LD; (b) youth with severe LD will show more incidents of school-related problems after their first involvement (e.g., attendance problems, disciplinary incidents such as in-school and out-of-school suspensions and expulsions) than youth without LD; (c) youth with severe LD who had school-related problems prior to their first JJ involvement will be at higher risk of recidivism than youth without LD; (d) lower levels of reading achievement will be associated with shorter periods of time to repeated offending; and (e) participation in the intervention will significantly decrease recidivism risk compared to other youth with severe LD who did not participate in the intervention.

Intervention:

The intervention component seeks to address three objectives: (1) to improve the reading skills of an understudied, high-risk population (JJ-involved youth) using an educational therapy that has been specifically designed for JJ-involved youth, provided in a 1:1 setting, and expanded with technology, including material relevant to daily living skills and appropriate reinforcement that will extend the program into the post-release period; (2) to reinforce skills and maintain reading gains made during the educational therapy, and increase the automaticity of skill use by using a high-interest "gamified" learning tool that youth will play on a SmartPhone given to them when they leave detention; and (3) to investigate the individual response to therapy with respect to other variables (e.g., attention, executive functioning, impulse control, learning ability, other academic achievement) collected at baseline.

Hypotheses. The key hypotheses of the intervention component seek to identify the factors associated with response to therapy for severe LD relative to pre-therapy functioning. We hypothesize that (a) overall improvement in reading will be related to pre-therapy academic skills, attention, and executive functioning; (b) inclusion of a metacognitive component in the therapy will provide carry-over effects, improving other academic skills; and (c) the gamification of the learning tool will result in robust technology usage, with a dose-response relationship between time spent on task and improvement in skills trained (and measured) via game play.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 14 and 16
* Conversational English ability (sufficient to benefit from the intervention program) based on the CASL-2 core score
* Reading below the 3rd grade level on the KTEA-3 pseudoword decoding subtest and the TOWRE-2 phonemic decoding efficiency subtest
* IQ at or above 70 on the KABC-II

Exclusion Criteria:

* Hearing or vision problem that would preclude the use of visual and auditory materials
* Developmental delay, autism spectrum disorder, or intellectual disability
* Known genetic syndrome
* Neurological disorder (e.g., epilepsy)
* Current psychosis or suicidal ideation
* Recent (within 6 months) traumatic brain injury

Ages: 14 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Reading Skills from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  Reading skills will be measured as a composite of two subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3):
  1. Letter & Word Recognition
  2. Reading Comprehension
  This standard score will be obtained based on the sum of subtest standard scores according to published norms.
Change in Decoding Skills from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  Decoding skills will be measured as a composite of two subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3):
  1. Letter & Word Recognition
  2. Nonsense Word Decoding
  This standard score will be obtained based on the sum of subtest standard scores according to published norms.
Change in Reading Understanding from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  Reading understanding will be measured as a composite of two subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3):
  1. Reading Comprehension
  2. Reading Vocabulary
  This standard score will be obtained based on the sum of subtest standard scores according to published norms.
Change in Comprehension from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  Comprehension will be measured as a composite of two subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3):
  1. Reading Comprehension
  2. Listening Comprehension
  This standard score will be obtained based on the sum of subtest standard scores according to published norms.
Change in Reading Fluency from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  The Test of Reading Efficiency, Second Edition (TOWRE-2) will be used to measure an individual's ability to pronounce printed words and phonemically regular nonwords accurately and fluently. Standard scores will be obtained according to published norms.
Change in Other Academic Skills from pre-intervention (baseline) to the week after intervention | Assessment of change will take place at pre-intervention (baseline), the week before intervention, after four weeks of intervention, and the week after intervention.
  Other academic skills will be measured as a composite of remaining subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3) and Woodcock-Johnson-IV Tests of Academic Achievement (WJ-IV):
  1. KTEA-3 Math Concepts & Application
  2. KTEA-3 Math Fluency
  3. KTEA-3 Rapid Automatized Naming Letters
  4. KTEA-3 Spelling
  5. WJ-IV Science
  6. WJ-IV Social Studies
  7. WJ-IV Humanities
  This standard score will be obtained based on the z-score of the sum of subtest standard scores at pre-intervention.

SECONDARY OUTCOMES:
Recidivism within 1 year post-intervention | Within 1 year post-intervention
  Recidivism will be computed as a dichotomous variable (yes/no) indicating whether an individual committed an offense within 1 year after participating in the intervention.
Number of days to recidivism within 1 year post-intervention | Within 1 year post-intervention
  For individuals who recidivated within 1 year after participating in the intervention, the number of days until the first offense post-intervention will be computed.
Detention within 1 year post-intervention | Within 1 year post-intervention
  This secondary outcome will be computed as a dichotomous variable (yes/no) indicating whether an individual has been detained within 1 year after participating in the intervention.
Number of days to detention within 1 year post-intervention | Within 1 year post-intervention
  For individuals who were detained within 1 year after participating in the intervention, the number of days until the first detention post-intervention will be computed
Adjudication within 1 year post-intervention | Within 1 year post-intervention
  This secondary outcome will be computed as a dichotomous variable (yes/no) indicating whether an individual has been adjudicated within 1 year after participating in the intervention.
Number of days to adjudication within 1 year post-intervention | Within 1 year post-intervention
  For individuals who were adjudicated within 1 year after participating in the intervention, the number of days until the first adjudication post-intervention will be computed.

OTHER OUTCOMES:
Changes in decoding skills as assessed by a SmartPhone App | Participants will use the SmartPhone App over a 14-week game-play period. Data will be collected during game play.
  A SmartPhone App will be used to assess changes in decoding skills over a 14-week game-play period. Specifically, changes in decoding skills will be measured by tracking the level participants reach in the SmartPhone game. Level is determined by word frequency (a proxy for difficulty).
Changes in word reading automaticity as assessed by a SmartPhone App | Participants will use the SmartPhone App over a 14-week game-play period. Data will be collected during game play.
  A SmartPhone App will be used to assess changes in word reading automaticity over a 14-week game-play period. Specifically, word reading automaticity will be measured by tracking the speed at which participants are able to make decisions regarding spellings and sounds of words presented during the SmartPhone game
Changes in breadth of vocabulary as assessed by a SmartPhone App | Participants will use the SmartPhone App over a 14-week game-play period. Data will be collected during game play.
  A SmartPhone App will be used to assess changes in breadth of vocabulary over a 14-week game-play period. Specifically, vocabulary will be measured by tracking the percent correct participants reach on vocabulary tasks in the SmartPhone game.

CONTACTS AND LOCATIONS:
Overall Officials: Elena L Grigorenko, PhD, Principal Investigator — BCM
Locations (1):
- Burnett-Bayland Rehabilitation Center (BBRC), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigorenko EL. Learning disabilities in juvenile offenders. Child Adolesc Psychiatr Clin N Am. 2006 Apr;15(2):353-71, viii. doi: 10.1016/j.chc.2005.11.001. PMID 16527660
- [Background] Archwamety, T. & Katsiyannis, A. Academic remediation, parole violations, and recidivism rates among delinquent youths. Remedial and Special Education 21, 161-170 (2000).
- [Background] Walker, H. M. & Sprague, J. R. The path to school failure, delinquency, and violence: Causal factors and some potential solutions. Intervention in School and Clinic 35, 67-73 (1999).
- [Background] Edmonds MS, Vaughn S, Wexler J, Reutebuch C, Cable A, Tackett KK, Schnakenberg JW. A Synthesis of Reading Interventions and Effects on Reading Comprehension Outcomes for Older Struggling Readers. Rev Educ Res. 2009 Mar 1;79(1):262-300. doi: 10.3102/0034654308325998. PMID 20072704
- [Background] Wexler, J., Pyle, N., Flower, A., Williams, J. L. & Cole, H. A synthesis of academic interventions for incarcerated adolescents. Review of Educational Research 84, 3-46 (2014).
- [Background] U.S. Department of Education, O. o. E. T. Enhancing teaching and learning through educational data mining and learning analytics: An issue brief. (U.S. Department of Education, Washington, DC, 2012)
- [Background] Baker, R. S. J. D. & Yacef, K. The state of educational data mining in 2009: A review and future visions. Journal of Educational Data Mining 1, 3-16 (2009).
- See also: Stevenson Learning Skills — http://www.stevensonlearning.com/